CLINICAL TRIAL: NCT00002711
Title: A PHASE I TRIAL OF COMBINED MODALITY THERAPY FOR LOCALIZED ESOPHAGEAL CANCER: CISPLATIN-PACLITAXEL FOLLOWED BY RADIATION THERAPY WITH CONCURRENT CISPLATIN AND ESCALATING DOSES OF PACLITAXEL
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Cancer of the Esophagus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 95-073; CDR0000064528 (Registry Identifier: PDQ (Physician Data Query)); NCI-H95-0791
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; recurrent esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Drug Therapy; Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: chemotherapy
Drug: cisplatin
Drug: paclitaxel
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy and radiation therapy in treating patients with cancer of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the maximum tolerated dose and recommend a phase II dose for paclitaxel (TAX) when administered as a 96-hour intravenous infusion with a weekly fixed dose of intravenous cisplatin (CDDP) during concurrent radiotherapy for patients with localized esophageal cancer. II. Estimate the response rate of patients treated with 2 courses of TAX/CDDP induction chemotherapy and the complete response rate of patients treated with TAX/CDDP and concurrent radiotherapy. III. Describe the toxic effects of TAX/CDDP prior to and during radiotherapy. IV. Describe the pharmacokinetics of TAX as a continuous infusion (CI) over 96 hours. V. Evaluate, by flow cytometry, the ability of CI TAX to block esophageal cancer cells in the G2-M phase of the cell cycle.

OUTLINE: After the MTD of TAX is reached on Part A, new patients are entered on Part B. The following acronyms are used: CDDP Cisplatin, NSC-119875 EBRT External-beam radiotherapy TAX Paclitaxel (Bristol-Myers), NSC-125973 PART A: Radiotherapy plus 2-Drug Combination Chemotherapy. EBRT using megavoltage equipment (>/= 10 MV recommended; electron boost allowed for subclavicular fossae); plus TAX/CDDP. PART B: 2-Drug Combination Induction Chemotherapy followed by Radiotherapy plus 2-Drug Combination Chemotherapy. TAX/CDDP; followed by EBRT as in Part A; plus TAX/CDDP.

PROJECTED ACCRUAL: At least 3 patients/dose will be entered on Part A (up to 24 patients) and 3-6 patients on Part B.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed epidermoid carcinoma or adenocarcinoma of the esophagus eligible for potentially curative radiotherapy Disease in one of the following categories: Newly diagnosed Locoregional failure after prior resection with curative intent Positive microscopic margin after palliative resection of all gross disease Disease clinically limited to esophagus T 1-4, any N, M0 Gastroesophageal junction tumor allowed No positive pleural, pericardial, or peritoneal cytology No tracheobronchial invasion on bronchoscopy, including tracheoesophageal fistula

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Hematopoietic: WBC more than 4,000/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 65 mL/min per 1.73 square meters Cardiovascular: No NYHA class 3/4 status No cerebral vascular disease No hypertension Other: No severe uncontrolled diabetes No uncontrolled infection No other medical condition that precludes treatment No mental status abnormality that precludes comprehension of or compliance with treatment No active cancer arising at another primary site other than basal cell carcinoma of the skin or in situ cervical carcinoma

PRIOR CONCURRENT THERAPY: No prior chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1995-10; Primary Completion 2000-10 (Actual); Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Paul Kelsen, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States